CLINICAL TRIAL: NCT06866223
Title: Emergent Bilinguals: the Relationship Between Child Language Proficiency and Language of Treatment on the Outcomes Children with Developmental Language Disorder
Brief Title: Emergent Bilinguals: Child Language Proficiency and Language of Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01DC020183 (NIH); STUDY00002073 (Other: University of Houston)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Developmental Language Disorder; Language Impairment
MeSH Terms: conditions — Language Development Disorders; Language Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two conditions: monolingual recast therapy delivered in English or Spanish, and interleaved therpay (bilingual therapy) Schools are randomly assigned to first treatment target (conditional adverbial clause; complement clause). The investigators use a cross-over design such that all children eventually receive treatment for all targets. Pretesting will be completed for both targets in both languages. Children will be stratified based on bilingual proficiency (Spanish-dominant (receptive English or simple sentences in English), English-dominant, Balanced) and randomly assigned to language of intervention. Children will receive 16 hours of recast therapy. After, both structures will be tested in both languages again. Then, treatment target will switch and children will receive an additional 16 hours of treatment for the second structure. At post-test, both structures will be tested in both languages.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monolingual therapy (Experimental): A trained, bilingual SLP will treat the targeted structure at a rate of ~ 1 recast per minute, for 16 hours spread over 9 weeks to obtain a planned dose of 912-1008 recasts (960 +/- 5%). Following evidence on enhanced conversational recasting, the SLP will obtain the child's attention before recasting and systematically vary the lexical items in the recasts. Children receiving monolingual Spanish therapy will have the entire treatment session conducted in the dominant language of the child (Spanish or English).
  Interventions: Behavioral: Sentence recast
- Interleaved therapy (Experimental): A trained, bilingual SLP will treat the targeted structure at a rate of ~ 1 recast per minute, for 16 hours spread over 9 weeks to obtain a planned dose of 912-1008 recasts (960 +/- 5%). Following evidence on enhanced conversational recasting, the SLP will obtain the child's attention before recasting and systematically vary the lexical items in the recasts. Children will receive therapy in the dominant language (Spanish or English) and will also be offered the opportunity to use the non-dominant language (Spanish or English) via communication bid in the child's non-dominant language every 3-5 minutes and continue in that language as long as the child responds. If the child does not respond or responds in their dominant language, the examiner will switch to the other language.
  Interventions: Behavioral: Sentence recast

INTERVENTIONS:
Behavioral: Sentence recast — Recast therapy is a well-established treatment for grammar in children with DLD. In this treatment, the adult repeats the child's own utterance, altering it to include the taught structure. It yields consistent large effect sizes (Hedge's g = 0.7-1.0) when focused on a single target and provided at a high dose (10-20 hrs. of therapy at a rate of ~1 recast/minute or ~600-1000 recasts total) for both morphology and syntax

SUMMARY:
Of the 12 million children in the USA growing up bilingual, about 1 million experience Developmental Language Disorder (DLD), a disorder in language learning and use. Currently there is no guidance for speech language pathologists (SLPs) as to the language of intervention for emergent Spanish-English bilingual children with DLD. This project will examine the relationship between language proficiency and the language of intervention, considering monolingual intervention (Spanish or English) and interleaved Spanish-English intervention with the goal of improving language outcomes and thereby strengthening long-term academic achievement

DETAILED DESCRIPTION:
More than 8.5 million children in the USA speak Spanish at home (U.S. Census Table S1601, 2020) with about a half million experiencing Developmental Language Disorder (DLD), a disorder in language learning and use not attributed to limited language exposure, autism, intellectual disability, etc. (Norbury et al., 2016). Bilingual children with DLD experience language-learning difficulties in both languages, including documented difficulty with complex syntax (Gutiérrez-Clellen, 1998; Jasso et al., under review). While it is self-evident that a monolingual child should be treated in their first language, currently there is no guidance for speech-language pathologists as to the language of intervention for bilingual children (Kohnert, et al., 2005). This is exacerbated by the fact that DLD varies in severity and bilingualism exists across a continuum, ranging from nearly monolingual in either language A or B to balanced bilingualism with good fluency in both languages. Furthermore, children who enter school with only limited proficiency in the majority language (e.g., English) rapidly become more proficient. This continuum is exemplified in our data. Recast therapy, an evidence-based intervention for grammatical difficulties (Cleave et al., 2015), is thought to work via mechanisms similar to priming (Leonard, 2011). Critically, cross-linguistic priming in bilingual children depends on proficiency (Vasilyeva et al., 2010) suggesting a need to align recast therapy with the child's proficiency profile (Gutiérrez-Clellen et al., 2012).

ELIGIBILITY:
Inclusion Criteria:

1. parent concerns and/or a history of receiving services in the public schools
2. age-specific cutoffs for the morphosyntax subtests for their best language (English or Spanish) on the Bilingual English Spanish Assessment. The cut-off score for best language for 4-year-olds is 84, for 5-year-olds is 85, and for 6-year-olds is 81.

   Using the best-language approach, these scores have a sensitivity over 90% and specificity over 80% for children between 4;0 and 6;11 years of age , which is considered acceptable for studies of diagnostic accuracy.
3. nonverbal IQ, as measured by the Kaufman Brief Intelligence Test-2, matrices subtest, will be at or above a standard score of 70.
4. pass a hearing screening test
5. participants must be emergent bilingual, that is children must be producing at least simple sentences in spontaneous speech in either Spanish or English and be exposed to both langauges
6. participants must be able to benefit from treatment for both conditional adverbial clauses and complement clauses, as evidenced by accuracy below 40% on 10-item elicited production probes in both languages

Exclusion Criteria:

1) children with significant sensory-motor concerns or psychiatric disorders per parent report will not be enrolled.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy on elicited production probes (conditional or nominal) | ~1 month before (Pre), 2 weeks before second structure (Mid) and 2 weeks after treatment (Post test)]
  Accuracy on elicited production probes are the primary outcome measure. There are 40 probes in total. Ten for Spanish conditionals, ten English conditionals, ten Spanish complement clauses and ten English complement clauses.

SECONDARY OUTCOMES:
Mean Length of Utterance and Subordination Index in English | ~1 month before (Pre), 2 weeks before second structure (Mid) and 2 weeks after treatment (Post test)]
  Calculated from a story retell in English. Mean length of utterance and subordination index.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
General summary data and individual-level data will be shared for the following variables: Age, parent education level, scores on standardized tests associated with eligibility and relative language proficiency, percent correct on pre-/mid-/post-test elicited production probes, and summary variables for language sample data (e.g., number of target utterances). This information will be made available in the form of a comma delimited text file and a code book. Individuals' identities by redacting birthdates and date of examination from the available records will be disguised by replacing names with coded alphanumeric values. Materials (books, probes, training tips, training videos, etc.) will be available to SLPs and other researchers upon request. Audio files cannot be fully deidentified; therefore, data at the child level will only be available with IRB approval.
  Supporting Information: